CLINICAL TRIAL: NCT02861807
Title: Mindfulness-Based Intervention and Transcranial Direct Current Brain Stimulation to Reduce Heavy Drinking: Efficacy and Mechanisms of Change
Brief Title: Mindfulness-Based Intervention and Transcranial Direct Current Brain Stimulation to Reduce Heavy Drinking
Acronym: MBItDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04316; R21AA024926 (NIH)
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-11

CONDITIONS: Alcohol Drinking; Alcohol Intoxication; Alcoholism
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active stimulation with mindfulness (Experimental): Brain stimulation with mindfulness-based relapse prevention. Treatment sessions will be 2 hours for 8 sessions, with the first 30 minutes consisting of transcranial direct current stimulation (tDCS) with the current set to 2.0 milliamps (mA) and guided meditation practice.
  Interventions: Device: Brain stimulation with mindfulness-based relapse prevention
- Sham brain stimulation with mindfulness (Sham Comparator): Brain stimulation with mindfulness-based relapse prevention. Treatment sessions will be 2 hours for 8 sessions, with the first 30 minutes consisting of transcranial direct current stimulation (tDCS) with the current set to ramp up to 2.0 milliamps (mA) and then ramp down to 0.0 mA and guided meditation practice.
  Interventions: Device: Brain stimulation with mindfulness-based relapse prevention

INTERVENTIONS:
Device: Brain stimulation with mindfulness-based relapse prevention — Participants will participate in weekly or twice weekly group mindfulness based relapse prevention (MBRP) + transcranial direct current stimulation (tDCS) intervention sessions for up to eight weeks. All participants will receive 8 two hour sessions of MBRP + tDCS, regardless of the group schedule. Subjects will receive 30 minutes of either active or sham tDCS stimulation, depending on their group assignment. After tDCS, sessions will include discussions of mindfulness as a means of coping with craving, cognitions, and emotions, role play exercises, and mindfulness practice.

SUMMARY:
Alcohol use disorder (AUD) impacts millions of Americans and is associated with significant behavioral, social, economic, medical, and neurobiological dysfunction, yet current behavioral treatments for AUD are only modestly effective. The proposed research will test the efficacy of a novel behavioral intervention, which combines brain stimulation with mindfulness-based relapse prevention, and is hypothesized to improve neural dysfunction and ultimately lead to large effect size reductions in heavy drinking among individuals with AUD. Given that mindfulness and brain stimulation are already available for "home use" there is great potential for the ultimate dissemination of the intervention on a large scale, which could have a significant impact on public health.

DETAILED DESCRIPTION:
Heavy drinking (defined as 4+/5+ drinks per occasion for women/men) and alcohol use disorder (AUD) are a significant public health problem. Modestly effective pharmacological and psychosocial treatments for AUD exist, yet some heavy drinking (i.e., relapse) is the most common outcome following AUD treatment. Continued development of innovative and efficacious interventions that reduce heavy drinking and specifically target risk factors for heavy drinking is thus clearly warranted. One novel intervention that has considerable promise for reducing heavy drinking is mindfulness-based relapse prevention (MBRP). MBRP is a behavioral intervention for substance use disorder that was designed to target experiences of craving and other risk factors for heavy drinking. Based on the results of numerous studies, MBRP is feasible and efficacious in the treatment of AUD. However the effect sizes of MBRP remain small and many individuals struggle with engaging in the mindfulness practices early in treatment. There is preliminary evidence that combining a non-invasive form of brain stimulation, transcranial direct current stimulation (tDCS), may improve engagement with mindfulness practices and lead to significant reductions in heavy drinking following treatment. The goal of the proposed study is to examine the efficacy of a mindfulness + tDCS intervention in reducing heavy drinking and impacting hypothesized mechanisms of behavior change among individuals with AUD who are interested in reducing their heavy drinking. In the proposed study, a research team with complementary expertise in AUD treatment, mindfulness-based interventions, brain stimulation, and cognitive neuroscience will combine self-report, behavioral, and neurophysiological data collection via electroencephalography (EEG) to study the psychological and neurophysiological mechanisms of treatment efficacy following a novel, promising intervention that combines brain stimulation with mindfulness training. The mindfulness based intervention in combination with active tDCS is hypothesized to lead to significant reductions in drinks per drinking day after 8 weeks of treatment and these reductions will be maintained up to 2 months following treatment. Further, the effect of active tDCS on drinks per drinking day at the 2 month follow-up will be mediated by greater mindfulness, greater inhibitory control and reductions in craving and negative affect during treatment and at the post-treatment assessment. Approximately 86 individuals meeting criteria for AUD will be randomly assigned to 8 sessions of either MBRP combined with active tDCS (up to 2.0 milliamp current) or MBRP combined with a sham tDCS (no current) control condition. The proposed study will examine the efficacy (Primary Aim) and psychological and neurophysiological mechanisms of treatment efficacy using behavioral measures and EEG (Secondary Aim). In addition to addressing the question of whether adding active tDCS to MBRP enhances efficacy, it will further examine issues of neurophysiological and behavioral treatment mechanisms to better inform the design of a future large efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

1. interested in reducing alcohol drinking
2. right-handed

Exclusion Criteria:

1. lifetime diagnosis of schizophrenia or bipolar disorder or current substance use disorder other than nicotine or marijuana
2. cardiac pacemaker
3. implantable defibrillator
4. metal objects in upper body that might interfere with tDCS, or that tDCS may interfere with their function, including metal plates, screws and prosthetics in head, certain older tattoos and permanent makeup using metal containing inks, aneurysm clips, neural stimulators of any kind, ear implants, insulin pumps, drug infusion devices and dental appliances
5. for females, pregnant or attempting to get pregnant
6. history of seizures or seizure disorder
7. allergic to latex, rubber, conductive medium like saline or electrode gel
8. if assigned to active tDCS and unable to tolerate 1.5 mA of tDCS during a baseline stimulation session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Psychology Clinical Neuroscience Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the data publicly available given that it will be a unique data set that will not only allow for further exploration by alcohol researchers, but also allow for methods development by the broader research community. The investigators plan to release the data to the public once the primary manuscripts describing the main findings of the study have been accepted for publication. Anonymized and preprocessed EEG data as well as deidentified behavioral and questionnaire data will be shared with investigators from institutions with a Federal Wide Assurance; all investigators with whom the data is shared will be included in the annual progress report. To ensure accessibility of the data set, instructions for obtaining the data set will be included in publications of the data collected under this grant.

REFERENCES:
- [Result] Witkiewitz K, Stein ER, Votaw VR, Wilson AD, Roos CR, Gallegos SJ, Clark VP, Claus ED. Mindfulness-Based Relapse Prevention and Transcranial Direct Current Stimulation to Reduce Heavy Drinking: A Double-Blind Sham-Controlled Randomized Trial. Alcohol Clin Exp Res. 2019 Jun;43(6):1296-1307. doi: 10.1111/acer.14053. Epub 2019 May 9. PMID 30977904
- [Result] Brown DR, Jackson TCJ, Claus ED, Votaw VR, Stein ER, Robinson CSH, Wilson AD, Brandt E, Fratzke V, Clark VP, Witkiewitz K. Decreases in the Late Positive Potential to Alcohol Images Among Alcohol Treatment Seekers Following Mindfulness-Based Relapse Prevention. Alcohol Alcohol. 2020 Feb 7;55(1):78-85. doi: 10.1093/alcalc/agz096. PMID 31825472
- [Derived] Gibson BC, Votaw VR, Stein ER, Clark VP, Claus E, Witkiewitz K. Transcranial Direct Current Stimulation Provides no Additional Benefit to Improvements in Self-Reported Craving Following Mindfulness-Based Relapse Prevention. Mindfulness (N Y). 2022 Jan;13(1):92-103. doi: 10.1007/s12671-021-01768-5. Epub 2021 Nov 26. PMID 35833199
- See also: Mindfulness recordings used for home practice during trial — https://abqresearch.org/mindfulness-recordings/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness
Started | 47 | 37
Attended Post-treatment Assessment | 34 | 18
Attended 2-month Follow-up | 32 | 20
Completed | 35 | 23
Not Completed | 12 | 14
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrawal by Subject | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness | Total
Number analyzed (Participants) | 47 | 37 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 33 | 74
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.43 (14.19) | 53.35 (11.41) | 52.27 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 28 | 22 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 31 | 21 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 32 | 22 | 54
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 47 | 37 | 84
Drinks per Drinking Occasion [Mean (Standard Deviation); unit: drinks per drinking occasion] — This measure, evaluating participants' number of drinks (standard drinks,14 grams of pure alcohol) per drinking occasion, was collected during the phone screen questionnaire, which occurred prior to the baseline assessment. Randomization to treatment condition was stratified based on this measure.
  drinks per drinking occasion | 6.64 (3.54) | 6.92 (4.35) | 6.76 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Drinking Day
Description: The Form 90 will be used to derive estimates of the primary outcome: drinks (standard drink=14 grams of pure alcohol) per drinking day.
Time Frame: Post-treatment and 2-month follow-up
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness
Number analyzed (Participants) | 35 | 23
drinks per drinking day
  Post-treatment assessment | 5.12 (3.14) | 5.64 (4.06)
  2-month follow-up | 4.95 (3.18) | 5.48 (4.28)

2. Secondary Outcome: Percent Heavy Drinking Days
Description: The Form 90 will be used to derive estimates of the secondary outcome: percent heavy drinking days, where heavy drinking is defined as 4+ drinks per occasion for women and 5+ drinks per occasion for men.
Time Frame: Post-treatment and 2-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness
Number analyzed (Participants) | 35 | 23
percentage of heavy drinking days
  Post-treatment assessment | 27.42 (30.54) | 25.93 (26.82)
  2-month follow-up | 29.51 (31.15) | 28.80 (33.16)

3. Other Pre Specified Outcome: Cue Reactivity at the Post-Treatment Assessment
Description: To measure cue reactivity to alcohol, the investigators will use a visual cue presentation task. Participants will view pictures of alcohol containing beverages and neutral pictures from the International Affective Pictures Series (IAPS)118 and from the web. Alcohol and neutral pictures will be matched for color and complexity as well as other potentially important confounds (e.g., presence of people). The investigators will examine responses to approximately 100 trials each of alcohol pictures and control pictures in a mixed event design (~15 minutes), in order to reduce predictability of the picture type. After viewing pictures participants reported craving for alcohol on a scale from 1 to 9 (1=no craving, 9=extreme craving) with higher scores indicating worse outcomes.
Time Frame: Post-treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness
Number analyzed (Participants) | 24 | 13
Score on a scale | 3.49 (1.81) | 3.06 (1.61)

4. Other Pre Specified Outcome: Reductions in Self-reported Craving
Description: Self-reported craving will be measured using the Penn Alcohol Craving Scale (scaled from 0 to 5 with higher scores indicate worse outcome = more craving) with higher scores mean a worse outcome.
Time Frame: 2 months following treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness
Number analyzed (Participants) | 32 | 20
Score on a scale | 2.24 (1.21) | 2.40 (1.42)

5. Other Pre Specified Outcome: Improvements in Inhibitory Control
Description: To examine inhibitory control, the investigators will use a Stop Signal Task in which participants make left-right judgments of the directionality of an arrow presented on the screen. For each trial, a circle will appear for 500 ms, followed by a left or right-pointing arrow for up to 1 second and between 500 ms and 2500 ms jittered inter-trial interval to reduce anticipatory responses. Approximately 25% of trials will be "stop trials" with a tone played to signal participants to inhibit the current response. This timing of the tone is dynamically adjusted to ensure successful inhibition on approximately 50% of trials. There will be 240 trials across 6 blocks (~10 minutes). Inhibitory control is measured by stop signal reaction time.
Time Frame: Post-treatment
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness
Number analyzed (Participants) | 28 | 15
milliseconds | 284.43 (94.85) | 266.06 (51.07)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Arm/Group | Active Stimulation With Mindfulness | Sham Brain Stimulation With Mindfulness
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/37
Other Adverse Events (participants affected / at risk) | 0/47 | 0/37

LIMITATIONS AND CAVEATS:
We were unable to assess alcohol biomarkers and relied entirely on self-reported drinking, which may be prone to errors. Another potential limitation is the relatively higher age and wide age range of this sample (52.3 years, SD 13.00, range 19-77).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT02861807/Prot_SAP_000.pdf